CLINICAL TRIAL: NCT02255435
Title: A Phase 2 Study of the Safety, Efficacy, and Pharmacodynamics of RTA 408 in the Treatment of Friedreich's Ataxia (MOXIe)
Brief Title: A Study to Learn About the Effects and Safety of RTA 408 (Omaveloxolone) in People Aged 16 to 40 With Friedreich's Ataxia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: AbbVie (Industry); Friedreich's Ataxia Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RTA 408-C-1402; 2024-517436-22 (Other: EU CTIS Number)
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Results first posted 2022-11-29 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Friedreich Ataxia
Keywords: RTA 408; RTA 408 Capsules; Oxidative Stress; Mitochondrial dysfunction; omaveloxolone
MeSH Terms: conditions — Friedreich Ataxia; Mitochondrial Diseases | interventions — omaveloxolone; ORF 50 transactivator

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Part 1 Omaveloxolone Capsules 2.5 and 5 mg (Experimental): omaveloxolone (RTA 408) Capsules, 2.5 mg administered orally one daily for 2 weeks, then 5 mg taken orally once daily for 10 weeks
  Interventions: Drug: Omaveloxolone Capsules, 2.5 mg; Drug: Omaveloxolone Capsules, 5 mg
- Part 1 Omaveloxolone Capsules 10 mg (Experimental): omaveloxolone (RTA 408) Capsules, 10 mg administered orally once daily for 12 weeks
  Interventions: Drug: Omaveloxolone Capsules, 10 mg
- Part 1 Omaveloxolone Capsules 20 mg (Experimental): Omaveloxolone (RTA 408) Capsules, 20 mg administered orally once daily for 12 weeks
  Interventions: Drug: Omaveloxolone Capsules, 20 mg
- Part 1 Omaveloxolone Capsules 40 mg (Experimental): Omaveloxolone (RTA 408) Capsules, 40 mg administered orally once daily for 12 weeks
  Interventions: Drug: Omaveloxolone Capsules, 40 mg
- Part 1 Omaveloxolone Capsules 80 mg (Experimental): Omaveloxolone (RTA 408) Capsules, 80 mg administered orally once daily for 12 weeks
  Interventions: Drug: Omaveloxolone Capsules, 80 mg
- Part 1 Omaveloxolone Capsules 160 mg (Experimental): Omaveloxolone (RTA 408) Capsules, 160 mg administered orally once daily for 12 weeks
  Interventions: Drug: Omaveloxolone Capsules, 160 mg
- Part 1 Omaveloxolone Capsules 300 mg (Experimental): Omaveloxolone (RTA 408) Capsules, 300 mg administered orally once daily for 12 weeks
  Interventions: Drug: Omaveloxolone Capsules, 300 mg
- Part 1 Placebo Capsules (Placebo Comparator): Placebo capsules administered orally once daily for 12 weeks
  Interventions: Drug: Placebo
- Part 2 Placebo Capsules (Placebo Comparator): Placebo capsules administered orally once daily for 48 weeks
  Interventions: Drug: Placebo
- Part 2 Omaveloxolone Capsules 150 mg (Experimental): Omaveloxolone (RTA 408) Capsules, 150 mg administered orally once daily for 48 weeks
  Interventions: Drug: Omaveloxolone Capsules, 150 mg

INTERVENTIONS:
Drug: Omaveloxolone Capsules, 2.5 mg
  Other Names: RTA 408 Capsules 2.5 mg
  Arms: Part 1 Omaveloxolone Capsules 2.5 and 5 mg
Drug: Omaveloxolone Capsules, 5 mg
  Other Names: RTA 408 capsules, 5 mg
  Arms: Part 1 Omaveloxolone Capsules 2.5 and 5 mg
Drug: Omaveloxolone Capsules, 10 mg
  Other Names: RTA 408 capsules, 10 mg
  Arms: Part 1 Omaveloxolone Capsules 10 mg
Drug: Placebo
  Arms: Part 1 Placebo Capsules; Part 2 Placebo Capsules
Drug: Omaveloxolone Capsules, 20 mg
  Other Names: RTA 408 capsules, 20 mg
  Arms: Part 1 Omaveloxolone Capsules 20 mg
Drug: Omaveloxolone Capsules, 40 mg
  Other Names: RTA 408 capsules, 40 mg
  Arms: Part 1 Omaveloxolone Capsules 40 mg
Drug: Omaveloxolone Capsules, 80 mg
  Other Names: RTA 408 capsules, 80 mg
  Arms: Part 1 Omaveloxolone Capsules 80 mg
Drug: Omaveloxolone Capsules, 160 mg
  Other Names: RTA 408 capsules, 160 mg
  Arms: Part 1 Omaveloxolone Capsules 160 mg
Drug: Omaveloxolone Capsules, 300 mg
  Other Names: RTA 408 capsules, 300 mg
  Arms: Part 1 Omaveloxolone Capsules 300 mg
Drug: Omaveloxolone Capsules, 150 mg
  Other Names: RTA 408 capsules, 150 mg
  Arms: Part 2 Omaveloxolone Capsules 150 mg

SUMMARY:
In this study, researchers are learning more about RTA 408, also known as omaveloxolone, BIIB141, or SKYCLARYS®. The main goal of this study is to learn more about the safety of RTA 408 and how it affects physical effort, movement, coordination, and how participants feel in daily life.

The main questions researchers want to answer in this study are:

* How much physical effort can a participant produce during a cycling test after 12 weeks of treatment?
* How do scores on the modified Friedreich's Ataxia Rating Scale (mFARS) change after 48 weeks?

Researchers will use the modified Friedreich's Ataxia Rating Scale (mFARS) to measure how FA affects the nervous system. The mFARS looks at movement ability, balance, coordination, speech, and how well the arms and legs work.

They will also use a cycling test to measure physical effort, along with questionnaires to learn how participants feel and function in daily life.

Safety will also be tested using physical exams, vital sign checks, echocardiograms (ECHO), electrocardiograms (ECG), and blood and urine tests.

The study will be done in 2 main parts, followed by an optional Extension period:

* In Part 1, participants will be randomly assigned to take different doses of RTA 408 or a placebo by mouth once a day for 12 weeks. A placebo looks like the study drug but contains no real medicine.
* Researchers will compare these doses to decide which one to use in Part 2.
* In Part 2, a different group of participants will take either the chosen dose of RTA 408 (150 mg) or placebo once a day for 48 weeks.
* Participants who complete Part 1 or Part 2 may be able to join an Extension period, where everyone receives RTA 408.
* In the Extension period, participants will continue to receive RTA 408 until the drug becomes commercially available or until they leave the study
* Participants in Part 1 will have up to 9 study visits and 2 phone calls. If they do not move onto the Extension period, they will stay in the study for up to 20 weeks.
* Participants in Part 2 will have up to 10 study visits and 3 phone calls. If they do not move onto the Extension period, they will stay in the study for up to 61 weeks.
* Participants in the Extension period will have 2 visits in the first month, followed by visits every 6 months.

DETAILED DESCRIPTION:
Friedreich's ataxia is an autosomal recessive cerebellar ataxia caused by triplet-repeat expansions. The causative mutation is a trinucleotide (GAA) repeat expansion in the first intron of the frataxin gene, leading to impaired transcription of frataxin. The pathological consequences of frataxin deficiency include a severe disruption of iron-sulfur cluster biosynthesis, mitochondrial iron overload coupled to cellular iron dysregulation, and an increased sensitivity to oxidative stress.

A hallmark of Friedreich's ataxia is impairment of antioxidative defense mechanisms, which play a major role in disease progression. Studies have demonstrated that nuclear factor erythroid-derived 2-related factor 2 (Nrf2) signaling is grossly impaired in participants with Friedreich's ataxia. Therefore, the ability of omaveloxolone (RTA 408) to activate Nrf2 and induce antioxidant target genes is hypothesized to be therapeutic in participants with Friedreich's ataxia.

This 2-part study will evaluate the efficacy, safety, and pharmacodynamics of omaveloxolone (RTA 408) in the treatment of participants with Friedreich's ataxia.

Part 1: The first part of this study will be a randomized, placebo-controlled, double-blind, dose-escalation study to evaluate the safety of omaveloxolone (RTA 408) at various doses in participants with Friedreich's ataxia.

Part 2: The second part of this study is a randomized, placebo-controlled, double-blind, parallel-group study to evaluate the safety and efficacy of omaveloxolone (RTA 408) 150 mg in participants with Friedreich's ataxia. Participants enrolled in Part 2 will be randomized 1:1 to receive omaveloxolone (RTA 408) 150 mg or placebo.

Extension: The extension will assess long-term safety and tolerability of omaveloxolone (RTA 408) in qualified participants with Friedreich's ataxia following completion of Part 1 or Part 2. Participants will not be unblinded to study treatment in Part 1 or Part 2 upon entering the extension study. Participants will receive open-label omaveloxolone (RTA 408) at 150 mg once daily.

ELIGIBILITY:
Inclusion Criteria:

1. Have genetically confirmed Friedreich's ataxia
2. Have a modified FARS score ≥20 and ≤80
3. Be male or female and ≥16 years of age and ≤40 years of age
4. Have no changes to exercise regimen within 30 days prior to Study Day 1 and be willing to remain on the same exercise regimen during the 16-week study period
5. Have the ability to complete maximal exercise testing
6. Be able to swallow capsules

Exclusion Criteria:

1. Have uncontrolled diabetes (HbA1c >11.0%)
2. Have B-type natriuretic peptide value >200 pg/mL
3. Have a history of clinically significant left-sided heart disease and/or clinically significant cardiac disease
4. Have known active fungal, bacterial, and/or viral infection, including human immunodeficiency virus or hepatitis virus (B or C)
5. Have known or suspected active drug or alcohol abuse
6. Have clinically significant abnormalities of clinical hematology or biochemistry, including but not limited to elevations greater than 1.5 times the upper limit of normal of aspartate aminotransferase, or alanine aminotransferase
7. Have any abnormal laboratory test value or serious pre-existing medical condition that, in the opinion of the investigator, would put the patient at risk by study enrollment
8. Have taken any of the following drugs within 7 days prior to Study Day 1 or plan to take any of these drugs during the time of study participation:

   1. Sensitive substrates for cytochrome P450 2C8 or 3A4 (e.g., repaglinide, midazolam, sildenafil)
   2. Moderate or strong inhibitors or inducers of cytochrome P450 3A4 (e.g., carbamazepine, phenytoin, ciprofloxacin, grapefruit juice)
   3. Substrates for p-glycoprotein transporter (e.g., ambrisentan, digoxin)
9. Have participated in any other interventional clinical study within 30 days prior to Study Day 1
10. Have a cognitive impairment that may preclude ability to comply with study procedures
11. Prior participation in a trial with omaveloxolone (RTA 408)

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 172 (Actual)
Dates: Start 2015-01-31 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2025-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (7):
  - UCLA, Los Angeles, California
  - University of Florida - Neurology, Gainesville, Florida
  - USF Ataxia Research Center, Tampa, Florida
  - Emory University Hospital - Neurology, Atlanta, Georgia
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - Ohio State University - Neurology, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Murdoch Childrens Research Institute, Parkville, Victoria, Australia
- Medical University Innsbruck, Innsbruck, Austria
- Neurological Institute Carlo Besta, Milan, Italy
- University College of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Lynch DR, Chin MP, Delatycki MB, Subramony SH, Corti M, Hoyle JC, Boesch S, Nachbauer W, Mariotti C, Mathews KD, Giunti P, Wilmot G, Zesiewicz T, Perlman S, Goldsberry A, O'Grady M, Meyer CJ. Safety and Efficacy of Omaveloxolone in Friedreich Ataxia (MOXIe Study). Ann Neurol. 2021 Feb;89(2):212-225. doi: 10.1002/ana.25934. Epub 2020 Nov 5. PMID 33068037
- [Derived] Lynch DR, Farmer J, Hauser L, Blair IA, Wang QQ, Mesaros C, Snyder N, Boesch S, Chin M, Delatycki MB, Giunti P, Goldsberry A, Hoyle C, McBride MG, Nachbauer W, O'Grady M, Perlman S, Subramony SH, Wilmot GR, Zesiewicz T, Meyer C. Safety, pharmacodynamics, and potential benefit of omaveloxolone in Friedreich ataxia. Ann Clin Transl Neurol. 2018 Nov 10;6(1):15-26. doi: 10.1002/acn3.660. eCollection 2019 Jan. PMID 30656180

RESULTS

PARTICIPANT FLOW:
Recruitment Details: MOXIe Part 1 and Part 2 were conducted under the same protocol. Participants enrolled in Part 1 were not allowed to enroll in Part 2. Patients with pes cavus were not to comprise more than 20% of all patients enrolled in Part 2.
Groups:
- Part 1 Omaveloxolone Capsules 2.5 and 5 mg: Omaveloxolone (RTA 408) Capsules, 2.5 mg administered orally one daily for 2 weeks, then 5 mg administered orally once daily for 10 weeks
  Omaveloxolone Capsules, 2.5 mg
  Omaveloxolone Capsules, 5 mg
- Part 1 Omaveloxolone Capsules 10 mg: Omaveloxolone (RTA 408) Capsules, 10 mg administered orally once daily for 12 weeks
  Omaveloxolone Capsules, 10 mg
- Part 1 Omaveloxolone Capsules 20 mg: Omaveloxolone (RTA 408) Capsules, 20 mg administered orally once daily for 12 weeks
  Omaveloxolone Capsules, 20 mg
- Part 1 Omaveloxolone Capsules 40 mg: Omaveloxolone (RTA 408) Capsules, 40 mg administered orally once daily for 12 weeks
  Omaveloxolone Capsules, 40 mg
- Part 1 Omaveloxolone Capsules 80 mg: Omaveloxolone (RTA 408) Capsules, 80 mg administered orally once daily for 12 weeks
  Omaveloxolone Capsules, 80 mg
- Part 1 Omaveloxolone Capsules 160 mg: Omaveloxolone (RTA 408) Capsules, 160 mg administered orally once daily for 12 weeks
  Omaveloxolone Capsules, 160 mg
- Part 1 Omaveloxolone Capsules 300 mg: Omaveloxolone (RTA 408) Capsules, 300 mg administered orally once daily for 12 weeks
  Omaveloxolone Capsules, 300 mg
- Part 1 Placebo Capsules: Placebo capsules administered orally once daily for 12 weeks
  Placebo
- Part 2 Placebo Capsules: Placebo capsules administered orally once daily for 48 weeks
  Placebo
- Part 2 Omaveloxolone Capsules 150 mg: Omaveloxolone (RTA 408) Capsules, 150 mg administered orally once daily for 48 weeks
  Omaveloxolone Capsules, 150 mg
Period: Overall Study
Arm/Group | Part 1 Omaveloxolone Capsules 2.5 and 5 mg | Part 1 Omaveloxolone Capsules 10 mg | Part 1 Omaveloxolone Capsules 20 mg | Part 1 Omaveloxolone Capsules 40 mg | Part 1 Omaveloxolone Capsules 80 mg | Part 1 Omaveloxolone Capsules 160 mg | Part 1 Omaveloxolone Capsules 300 mg | Part 1 Placebo Capsules | Part 2 Placebo Capsules | Part 2 Omaveloxolone Capsules 150 mg
Started | 6 | 6 | 6 | 6 | 6 | 12 | 10 | 17 | 52 | 51
Number of Participants With Pes Cavus | 2 | 2 | 3 | 2 | 2 | 8 | 3 | 10 | 10 | 10
Completed | 6 | 6 | 6 | 6 | 6 | 12 | 10 | 16 | 51 | 45
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 6
Not completed — Patient's Limited Time Availability | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Not completed — Administrative reasons | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized patients, whether or not they received study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Omaveloxolone Capsules 2.5 and 5 mg | Part 1 Omaveloxolone Capsules 10 mg | Part 1 Omaveloxolone Capsules 20 mg | Part 1 Omaveloxolone Capsules 40 mg | Part 1 Omaveloxolone Capsules 80 mg | Part 1 Omaveloxolone Capsules 160 mg | Part 1 Omaveloxolone Capsules 300 mg | Part 1 Placebo Capsules | Part 2 Placebo Capsules | Part 2 Omaveloxolone Capsules 150 mg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 12 | 10 | 17 | 52 | 51 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (5.98) | 25.5 (7.4) | 28.3 (6.8) | 27.7 (7.53) | 24.3 (4.8) | 25.3 (6.51) | 25.6 (7.24) | 24.4 (6.74) | 24.1 (7.85) | 23.4 (6.08) | 24.5 (6.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 1 | 3 | 5 | 5 | 10 | 17 | 31 | 85
  Male | 2 | 2 | 1 | 5 | 3 | 7 | 5 | 7 | 35 | 20 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 7
  Not Hispanic or Latino | 6 | 5 | 6 | 6 | 6 | 12 | 10 | 16 | 49 | 49 | 165
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 6 | 6 | 11 | 10 | 16 | 50 | 50 | 167
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 5
Region of Enrollment [Number; unit: participants]
  Austria | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 6 | 3 | 14
  United States | 6 | 6 | 6 | 6 | 5 | 8 | 7 | 16 | 35 | 36 | 131
  United Kingdom | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 8
  Italy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 7
  Australia | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 5 | 12
Peak Work [Mean (Standard Deviation); unit: W/kg] — Peak work attained during maximal exercise testing. Cycle ergometry using a recumbent stationary bicycle was used, and workload was increased incrementally. Peak work is defined as the workload at which patients reach maximal volition (defined as an inability to continue to exercise due to exhaustion).
  W/kg | 1.2 (0.696) | 0.78 (0.677) | 1.25 (0.838) | 0.72 (0.565) | 1.6 (0.556) | 1.18 (0.646) | 0.88 (0.521) | 0.99 (0.637) | 1.23 (0.622) | 1.09 (0.576) | 1.12 (0.621)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Peak Work (in Watts/kg) During Exercise Testing at Week 12 in Part 1
Description: Peak work attained during maximal exercise testing. Cycle ergometry using a recumbent stationary bicycle was used, and workload was increased incrementally. Peak work is defined as the workload at which patients reach maximal volition (defined as an inability to continue to exercise due to exhaustion).
Time Frame: Baseline through 12 weeks after participant receives the first dose in Part 1.
Population: All randomized patients in Part 1, whether or not they received study drug
Measure: Least Squares Mean (95% Confidence Interval); unit: W/kg
Arm/Group | Part 1 Omaveloxolone Capsules 2.5 and 5 mg | Part 1 Omaveloxolone Capsules 10 mg | Part 1 Omaveloxolone Capsules 20 mg | Part 1 Omaveloxolone Capsules 40 mg | Part 1 Omaveloxolone Capsules 80 mg | Part 1 Omaveloxolone Capsules 160 mg | Part 1 Omaveloxolone Capsules 300 mg | Part 1 Placebo Capsules
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 12 | 10 | 17
W/kg | 0.14 [0.02 to 0.26] | 0.07 [-0.05 to 0.18] | -0.09 [-0.20 to 0.03] | 0.06 [-0.06 to 0.18] | 0 [-0.11 to 0.12] | 0.02 [-0.06 to 0.10] | 0.07 [-0.02 to 0.17] | 0.04 [-0.03 to 0.11]
Statistical Analysis 1: Comparison: Part 1 Omaveloxolone Capsules 2.5 and 5 mg vs Part 1 Placebo Capsules; Test type: Superiority; p = 0.1524, Mixed Models Analysis; Treatment group, time, and the interaction between treatment and time were used as fixed factors; LS Mean difference (Net) = 0.10, 95% CI 2-sided [-0.04 to 0.23] — Difference is omaveloxolone - placebo
Statistical Analysis 2: Comparison: Part 1 Omaveloxolone Capsules 10 mg vs Part 1 Placebo Capsules; Test type: Superiority; p = 0.7086, Mixed Models Analysis; Treatment group, time, and the interaction between treatment and time were used as fixed factors; LS Mean difference (Net) = 0.03, 95% CI 2-sided [-0.11 to 0.16] — Difference is omaveloxolone - placebo
Statistical Analysis 3: Comparison: Part 1 Omaveloxolone Capsules 20 mg vs Part 1 Placebo Capsules; Test type: Superiority; p = 0.0651, Mixed Models Analysis; Treatment group, time, and the interaction between treatment and time were used as fixed factors; LS Mean difference (Net) = -0.13, 95% CI 2-sided [-0.26 to 0.01] — Difference is omaveloxolone - placebo
Statistical Analysis 4: Comparison: Part 1 Omaveloxolone Capsules 40 mg vs Part 1 Placebo Capsules; Test type: Superiority; p = 0.7937, Mixed Models Analysis; Treatment group, time, and the interaction between treatment and time were used as fixed factors; LS Mean difference (Net) = 0.02, 95% CI 2-sided [-0.12 to 0.15] — Difference is omaveloxolone - placebo
Statistical Analysis 5: Comparison: Part 1 Omaveloxolone Capsules 80 mg vs Part 1 Placebo Capsules; Test type: Superiority; p = 0.5587, Mixed Models Analysis; Treatment group, time, and the interaction between treatment and time were used as fixed factors; LS Mean difference (Net) = -0.04, 95% CI 2-sided [-0.18 to 0.10] — Difference is omaveloxolone - placebo
Statistical Analysis 6: Comparison: Part 1 Omaveloxolone Capsules 160 mg vs Part 1 Placebo Capsules; Test type: Superiority; p = 0.7285, Mixed Models Analysis; Treatment group, time, and the interaction between treatment and time were used as fixed factors; LS Mean difference (Net) = -0.02, 95% CI 2-sided [-0.13 to 0.09] — Difference is omaveloxolone - placebo
Statistical Analysis 7: Comparison: Part 1 Omaveloxolone Capsules 300 mg vs Part 1 Placebo Capsules; Test type: Superiority; p = 0.5802, Mixed Models Analysis; Treatment group, time, and the interaction between treatment and time were used as fixed factors; LS Mean difference (Net) = 0.03, 95% CI 2-sided [-0.09 to 0.15] — Difference is omaveloxolone - placebo
Statistical Analysis 8: Comparison: Part 1 Omaveloxolone Capsules 2.5 and 5 mg vs Part 1 Omaveloxolone Capsules 10 mg vs Part 1 Omaveloxolone Capsules 20 mg vs Part 1 Omaveloxolone Capsules 40 mg vs Part 1 Omaveloxolone Capsules 80 mg vs Part 1 Omaveloxolone Capsules 160 mg vs Part 1 Omaveloxolone Capsules 300 mg vs Part 1 Placebo Capsules; Comparison of Omaveloxolone capsules pooled with Placebo capsules; Test type: Superiority; p = 0.9698, Mixed Models Analysis; Treatment group, time, and the interaction between treatment and time were used as fixed factors; LS Mean difference (Net) = -0.00, 95% CI 2-sided [-0.08 to 0.08] — Difference is omaveloxolone - placebo

2. Primary Outcome: Change in the Modified Friedreich's Ataxia Rating Scale (mFARS) at Week 48 in Part 2
Description: The mFARS includes 4 of the 5 sections of the Friedreich's Ataxia Rating Scale (FARS): bulbar (score 0 to 11), upper limb coordination (score 0 to 36), lower limb coordination (score 0 to 16), and upright stability (score 0 to 36). The minimum score is 0 and the maximum score is 99. A lower score indicates better neurological function.
Time Frame: 48 weeks after participant receives the first dose in Part 2
Population: Full analysis set (all patients in Part 2 randomized without pes cavus who have at least one post-baseline measurement)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part 2 Placebo Capsules | Part 2 Omaveloxolone Capsules 150 mg
Number analyzed (Participants) | 42 | 40
score on a scale | 0.85 (0.640) | -1.55 (0.689)
Statistical Analysis 1: Comparison: Part 2 Placebo Capsules vs Part 2 Omaveloxolone Capsules 150 mg; Test type: Superiority; p = 0.0141, Mixed Models Analysis; Fixed factors: treatment group, time, interaction between treatment and time, interaction between baseline and time; covariates: site, baseline mFARS; LS Mean difference (Net) = -2.40, 95% CI 2-sided [-4.31 to -0.50], Standard Error of Mean 0.956 — Difference is omaveloxolone - placebo

3. Secondary Outcome: Change in the Modified Friedreich's Ataxia Rating Scale (mFARS) at Week 12 in Part 1
Description: as for outcome 2
Time Frame: 12 weeks after participant receives the first dose in Part 1
Population: All randomized patients in Part 1, whether or not they received study drug
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Part 1 Omaveloxolone Capsules 2.5 and 5 mg | Part 1 Omaveloxolone Capsules 10 mg | Part 1 Omaveloxolone Capsules 20 mg | Part 1 Omaveloxolone Capsules 40 mg | Part 1 Omaveloxolone Capsules 80 mg | Part 1 Omaveloxolone Capsules 160 mg | Part 1 Omaveloxolone Capsules 300 mg | Part 1 Placebo Capsules
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 12 | 10 | 17
score on a scale | -3.26 [-5.82 to -0.70] | -1.97 [-4.53 to 0.59] | -2.44 [-5.00 to 0.12] | -2.4 [-4.96 to 0.16] | -2.88 [-5.44 to -0.31] | -3.75 [-5.56 to -1.94] | -0.88 [-2.86 to 1.11] | -1.43 [-2.97 to 0.11]
Statistical Analysis 1: Comparison: Part 1 Omaveloxolone Capsules 2.5 and 5 mg vs Part 1 Placebo Capsules; Test type: Superiority; p = 0.2310, Mixed Models Analysis; Treatment group, time, and the interaction between treatment and time were used as fixed factors; LS Mean difference (Net) = -1.81, 95% CI 2-sided [-4.80 to 1.18] — Difference is omaveloxolone - placebo
Statistical Analysis 2: Comparison: Part 1 Omaveloxolone Capsules 10 mg vs Part 1 Placebo Capsules; Test type: Superiority; p = 0.7298, Mixed Models Analysis; Treatment group, time, and the interaction between treatment and time were used as fixed factors; LS Mean difference (Net) = -0.52, 95% CI 2-sided [-3.51 to 2.47] — Difference is omaveloxolone - placebo
Statistical Analysis 3: Comparison: Part 1 Omaveloxolone Capsules 20 mg vs Part 1 Placebo Capsules; Test type: Superiority; p = 0.5102, Mixed Models Analysis; Treatment group, time, and the interaction between treatment and time were used as fixed factors; LS Mean difference (Net) = -0.99, 95% CI 2-sided [-3.99 to 2.00] — Difference is omaveloxolone - placebo
Statistical Analysis 4: Comparison: Part 1 Omaveloxolone Capsules 40 mg vs Part 1 Placebo Capsules; Test type: Superiority; p = 0.5281, Mixed Models Analysis; Treatment group, time, and the interaction between treatment and time were used as fixed factors; LS Mean difference (Net) = -0.95, 95% CI 2-sided [-3.94 to 2.04] — Difference is omaveloxolone - placebo
Statistical Analysis 5: Comparison: Part 1 Omaveloxolone Capsules 80 mg vs Part 1 Placebo Capsules; Test type: Superiority; p = 0.3458, Mixed Models Analysis; Treatment group, time, and the interaction between treatment and time were used as fixed factors; LS Mean difference (Net) = -1.42, 95% CI 2-sided [-4.42 to 1.57] — Difference is omaveloxolone - placebo
Statistical Analysis 6: Comparison: Part 1 Omaveloxolone Capsules 160 mg vs Part 1 Placebo Capsules; Test type: Superiority; p = 0.0587, Mixed Models Analysis; Treatment group, time, and the interaction between treatment and time were used as fixed factors; LS Mean difference (Net) = -2.30, 95% CI 2-sided [-4.68 to 0.09] — Difference is omaveloxolone - placebo
Statistical Analysis 7: Comparison: Part 1 Omaveloxolone Capsules 300 mg vs Part 1 Placebo Capsules; Test type: Superiority; p = 0.6480, Mixed Models Analysis; Treatment group, time, and the interaction between treatment and time were used as fixed factors; LS Mean difference (Net) = 0.58, 95% CI 2-sided [-1.94 to 3.10] — Difference is omaveloxolone - placebo
Statistical Analysis 8: Comparison: Part 1 Omaveloxolone Capsules 2.5 and 5 mg vs Part 1 Omaveloxolone Capsules 10 mg vs Part 1 Omaveloxolone Capsules 20 mg vs Part 1 Omaveloxolone Capsules 40 mg vs Part 1 Omaveloxolone Capsules 80 mg vs Part 1 Omaveloxolone Capsules 160 mg vs Part 1 Omaveloxolone Capsules 300 mg vs Part 1 Placebo Capsules; Comparison of Omaveloxolone capsules pooled with Placebo capsules; Test type: Superiority; p = 0.2174, Mixed Models Analysis; Treatment group, time, and the interaction between treatment and time were used as fixed factors; LS Mean difference (Net) = -1.10, 95% CI 2-sided [-2.87 to 0.66] — Difference is omaveloxolone - placebo

ADVERSE EVENTS:
Time Frame: 16 weeks for Part 1 and 52 weeks for Part 2
Description: After the first dose, documentation of adverse events was to continue until 30 days following administration of the final dose of study medication, regardless of their relationship to study drug or their clinical significance.
Arm/Group | Part 1 Omaveloxolone Capsules 2.5 and 5 mg | Part 1 Omaveloxolone Capsules 10 mg | Part 1 Omaveloxolone Capsules 20 mg | Part 1 Omaveloxolone Capsules 40 mg | Part 1 Omaveloxolone Capsules 80 mg | Part 1 Omaveloxolone Capsules 160 mg | Part 1 Omaveloxolone Capsules 300 mg | Part 1 Placebo Capsules | Part 2 Placebo Capsules | Part 2 Omaveloxolone Capsules 150 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/10 | 0/17 | 0/52 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/10 | 2/17 | 3/52 | 5/51
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6 | 5/6 | 6/6 | 6/6 | 11/12 | 10/10 | 16/17 | 52/52 | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Omaveloxolone Capsules 2.5 and 5 mg (N=6) | Part 1 Omaveloxolone Capsules 10 mg (N=6) | Part 1 Omaveloxolone Capsules 20 mg (N=6) | Part 1 Omaveloxolone Capsules 40 mg (N=6) | Part 1 Omaveloxolone Capsules 80 mg (N=6) | Part 1 Omaveloxolone Capsules 160 mg (N=12) | Part 1 Omaveloxolone Capsules 300 mg (N=10) | Part 1 Placebo Capsules (N=17) | Part 2 Placebo Capsules (N=52) | Part 2 Omaveloxolone Capsules 150 mg (N=51)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Omaveloxolone Capsules 2.5 and 5 mg (N=6) | Part 1 Omaveloxolone Capsules 10 mg (N=6) | Part 1 Omaveloxolone Capsules 20 mg (N=6) | Part 1 Omaveloxolone Capsules 40 mg (N=6) | Part 1 Omaveloxolone Capsules 80 mg (N=6) | Part 1 Omaveloxolone Capsules 160 mg (N=12) | Part 1 Omaveloxolone Capsules 300 mg (N=10) | Part 1 Placebo Capsules (N=17) | Part 2 Placebo Capsules (N=52) | Part 2 Omaveloxolone Capsules 150 mg (N=51)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (4)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Friedreich's ataxia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 3 (3) | 11 (21)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 5 (6) | 10 (12)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 1 (1) | 7 (8) | 17 (22)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 8 (9)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Energy increased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 7 (7) | 11 (11)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 2 (2)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (11) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (8)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 9 (13) | 7 (7)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (4) | 1 (1) | 5 (5) | 2 (2) | 2 (3) | 4 (4) | 6 (10) | 1 (1) | 15 (29) | 14 (20)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 19 (43) | 17 (29)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 12 (21) | 13 (18)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 8 (10) | 8 (16)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 8 (12) | 5 (7)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (3)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 19 (20)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 11 (12)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (4)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 3 (4)
Glucose urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Very low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (6)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 10 (13) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (6) | 7 (9)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 8 (13)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (3) | 4 (4) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 3 (3) | 13 (35) | 19 (30)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Muscle spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 3 (3)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (7)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 9 (10)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (5):
  • Study Protocol: Main Protocol (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT02255435/Prot_000.pdf
  • Study Protocol: United Kingdom Protocol (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT02255435/Prot_001.pdf
  • Statistical Analysis Plan: Part 1 (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT02255435/SAP_002.pdf
  • Statistical Analysis Plan: Part 2 (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT02255435/SAP_003.pdf
  • Statistical Analysis Plan: Part 2 Addendum (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT02255435/SAP_004.pdf